CLINICAL TRIAL: NCT00441480
Title: Effect of Plant Sterols Esterified to Fish Oil Fatty Acids on Plasma Lipid Levels in Healthy, Hyperlipidemic Subjects
Brief Title: Effect of Plant Sterols Esterified to Fish Oil Fatty Acids on Plasma Lipid Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Enzymotec (Industry)
Responsible Party: Yael Herzog, Enzymotec LTD
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CardiaBeat_003
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2009-08-14 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Dyslipidemia
Keywords: Hypercholesterolemia; Hypertriglyceridemia; Plant sterol; Cholesterol; Fish oil
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plant sterol esters (Active Comparator): plant sterols esterified to fish oil fatty acids
  Interventions: Dietary Supplement: Plant sterols esters
- placebo (Placebo Comparator): Corn oil
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Plant sterols esters — 1.6g phytosterols and 1.3g omega-3 fatty acids per day
  Other Names: PS-FO
  Arms: Plant sterol esters
Dietary Supplement: placebo — 4 gr of corn oil
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether plant sterols esterified to fish oil fatty acids in a fish oil matrix improve the lipid profile, predominantly LDL-cholesterol and TG concentrations in healthy hyperlipidemic subjects.

DETAILED DESCRIPTION:
Phytosterols and omega-3 fatty acids (n-3) are natural food ingredients with potential cardiovascular (CVD) benefits. Phytosterols inhibit dietary cholesterol absorption and biliary cholesterol re-absorption, thereby reducing blood cholesterol levels, while consumption of n-3 is associated with a significant reduction in plasma triglyceride concentrations. Furthermore, n-3 may also beneficially modify a number of other risk factors of CHD, like anti-inflammatory and anti-thrombotic.

The primary objective of this study is to determine whether plant sterols esterified to fish oil fatty acids in a fish oil matrix improve the lipid profile, predominantly LDL-cholesterol and TG concentrations in healthy hyperlipidemic subjects. In addition the supplement efficacy to lower other CVD-related risk factors of healthy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years old and ≤ 70 years old, capable and willing to give written informed consent.
* Subject must have hyperlipidemia at the screening visit and at the end of the run-in period, defined as: fasting plasma triglycerides > 150 mg/dl and < 500 mg/dl, LDL-cholesterol > 130 mg/dl and < 190 mg/dl.
* Fasting plasma glucose (FPG) levels at the screening visit < 110 mg/dl.
* Female patient who is of reproductive potential agree to use acceptable methods of birth control
* Female patient who is currently receiving hormone replacement therapy continuously 12 weeks before visit 1 (on stable dose) and will agree to do so during the study.

Exclusion Criteria:

* Receiving medications or supplements known to affect lipid metabolism.
* Uncontrolled hypertension or thyroid disease.
* Consume unusual diets - will be determined at the discretion of the investigator.
* Gained or lost more than 3 kg during the run-in period.
* Patient has history of malignancy ≤ 5 years.
* Patients with clinical ischemic CV disease on treatment
* Consume 200 grams fish x 2 a week.
* Gastrointestinal disease or any disease that the investigator feels would compromise the patient safety or limit his/her successful participation to the study.
* Patient has type 1 or type 2 diabetes mellitus.
* Patient has uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Patient has had active peptic ulcer disease within 3 months of visit 1.
* Woman patient is pregnant or breast-feeding or expecting to conceive during the study.
* Patient has a history of hypersensitivity or allergy to fish, fish oil, corn oil or soy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Harats, M.D., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Bitzur R, Cohen H, Cohen T, Dror TW, Herzog Y, Lifshitz Y, Lubish T, Harats D, Rubinstein A. The metabolic effects of omega-3 plant sterol esters in mixed hyperlipidemic subjects. Cardiovasc Drugs Ther. 2010 Dec;24(5-6):429-37. doi: 10.1007/s10557-010-6249-5. PMID 20617456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period:r May 2007-Jan 2008 (8 months) Medical center
Pre-assignment Details: 10 -14 days run-in phase during which they received placebo capsules. Run-in phase enabled to exclude subjects who had an unstable weight (gained or lost more than 3 kg) during this period or who didn't meet entry criteria of LDL-c and TG at screening visit and at baseline visit.
Groups:
- PS-FO: plant sterols esterified to fish oil fatty acids
- Control: Corn oil
Period: Overall Study
Arm/Group | PS-FO | Control
Started | 46 | 45
Completed | 43 | 41
Not Completed | 3 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PS-FO | Control | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 43 | 84
  >=65 years | 5 | 2 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (10.8) | 49.4 (9.3) | 50.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 37 | 34 | 71
Region of Enrollment [Number; unit: participants]
  Israel | 46 | 45 | 91

OUTCOME MEASURES:

1. Primary Outcome: LDL Cholesterol
Description: Average of blood test results at -10 and 0 days (before and after run-in period)
Time Frame: at baseline
Population: Subjects whose body weight were changed from baseline value by more than 3 kg during the interventions or had compliance below 65% were excluded from analysis before breaking the randomization code. It was done since these changes may have a significant influence on the study end points
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 159.7 (17.22) | 157.8 (15.54)

2. Secondary Outcome: Triglycerides
Description: Average of blood test results at -10 and 0 weeks (before and after run-in period)
Time Frame: at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 244.9 (83.2) | 248.9 (65.4)

3. Secondary Outcome: Triglycerides
Description: Blood test results following 12 weeks of intervention
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 193.9 (77.0) | 233.0 (95.0)

4. Secondary Outcome: Total Cholesterol
Description: Average of blood test results at -10 and 0 weeks (before and after run-in period)
Time Frame: at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 244.3 (24.7) | 239.6 (22.7)

5. Secondary Outcome: Total Cholesterol
Description: Blood test results following 12 weeks of intervention
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 233.8 (28.0) | 236.5 (27.7)

6. Secondary Outcome: HDL Cholesterol
Description: Average of blood test results at -10 and 0 weeks (before and after run-in period)
Time Frame: at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 46.0 (9.1) | 44.2 (7.7)

7. Primary Outcome: LDL-C
Description: Blood test results following 12 weeks of intervention
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: md/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
md/dl | 154.7 (21.0) | 155.1 (20.1)

8. Secondary Outcome: HDL-cholestrol
Description: Blood test results following 12 weeks of intervention
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 46.4 (9.8) | 44.7 (10.5)

9. Secondary Outcome: CRP
Description: Blood test results on day 0 of High sensitivity C Reactive Protein
Time Frame: at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/l | 3.07 (3.45) | 3.25 (2.61)

10. Secondary Outcome: CRP
Description: Blood test results following 12 weeks of intervention of High sensetivity C reactive protein
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/l | 2.47 (2.45) | 4.51 (4.15)

11. Secondary Outcome: Apolipoprotein B100
Description: Blood test results on day 0
Time Frame: at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 130.6 (15.7) | 129.4 (14.3)

12. Secondary Outcome: Apolipoprotein B100
Description: Blood test results follwing 12 weeks of intervention
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 130.0 (19.1) | 130.3 (17.0)

13. Secondary Outcome: Apolipoprotein A
Description: Blood test on day 0
Time Frame: at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 126.3 (13.5) | 125.6 (13.6)

14. Secondary Outcome: Apolipoprotein A
Description: Blood test results following 12 weeks of intervention
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PS-FO | Control
Number analyzed (Participants) | 34 | 33
mg/dl | 128.2 (14.5) | 127.8 (16.3)

ADVERSE EVENTS:
Arm/Group | PS-FO | Control
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 1/46 | 1/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PS-FO (N=46) | Control (N=45)
abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Itching rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No